CLINICAL TRIAL: NCT06134427
Title: Body Fat Percentage Prediction Model of the Basic Combat Training Effect on Army Candidate' Body Composition in Indonesia
Brief Title: Body Fat Percentage Prediction Model After Basic Combat Training on Army Candidate in Indonesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Dwi Monik Purnamasari, Principal investigator, Indonesia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: Ket- 105/UN2.F10.D11/PPM.00.02
Record Dates: First submitted 2023-11-04; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Military Activity
Keywords: Anthropometry; body composition; basic combat training; predictive model formula; military cadets

STUDY DESIGN:
Intervention Model Description: Pre-Experimental Model One-Group Pretest-Posttest Design
Masking Description: statistical analyses using ID (not name) data set
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- basic combat training (Other): Pre experimental design, only one group with intervention basic combat training
  Interventions: Other: basic combat training (investigator did not design the intervention)

INTERVENTIONS:
Other: basic combat training (investigator did not design the intervention) — 12 weeks basic combat training is 12 weeks is a compulsory program for all cadets accepted in republic indonesia defense university

SUMMARY:
This research is a quantitative study using the Pre-Experimental Model One-Group Pretest-Posttest Design with total sampling from the Republic of Indonesia Defense University batch 4 cadets that fullfiled criteria. The intervention is 12 weeks basic combat training (only one group), a compulsory program for cadets.

DETAILED DESCRIPTION:
the purpose of this study is know the effect of basic combat training on the anthropometry and body fat percentage prediction model of army cadets after basic combat training in Indonesia

ELIGIBILITY:
Inclusion Criteria:

* Students as fourth batch in bachelor program in Indonesia Defense University
* Aged 16-18 years

Exclusion Criteria:

* Drop out or resign from Indonesia Defense University during research
* Having emergency condition during examination

Ages: 16 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — analyses of female and male subject were separated
Enrollment: 258 (Actual)
Dates: Start 2023-05-17 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Anthropometry after basic combat training in cadets of Indonesia | 12 weeks
  Pre post data of z score BMI for age based on who anhtroplus in standar deviation. Weight measured by BIA omron HBF 375, height measured by Microtoise OneMed. Height only measured once before combat training
Anthropometry after basic combat training in cadets of Indonesia | 12 weeks
  Pre post data of weight in measured by BIA omron HBF 375
Anthropometry after basic combat training in cadets of Indonesia | 12 weeks
  Pre post data of waist circumference in cm measured by non-elastic measuring tape OneMed OD 235.
Anthropometry after basic combat training in cadets of Indonesia | 12 weeks
  Pre post data of triceps skinfold, bicep skinfold, subscapular skinfold, suprailiac skinfold, and skinfold thickness (aggregate measurement of tricep, bicep, subscapular, and suprailiac skinfold) in mm measured by Harpenden Caliper
Body composition after basic combat training in cadets of Indonesia | 12 weeks
  Pre post data of body fat percentage in %, Whole body subcutaneous fat in %, whole body skeletal muscle in %, measured by BIA Omron type HBF 375
Body Fat Percentage Prediction Model of the Basic Combat Training (BCT) Effect on Army Candidate' | 12 weeks
  Total and delta predictive equation formula of body fat percentage after BCT based on variables delta and total value before bct of z score bmi for age, waist circumference, skinfold thickness, sleep quality measured by psqi, total daily carbohydrate, calorie, protein, fat intake based on semi quantitave food frequency questionnaires for macronutrient in bahasa Indonesia, and physical activity measured by IPAQ questionairres in bahasa indonesia. Variables body fat percentage before bct include as predictor in total body fat percentage prediction equation formula after BCT
Sleep quality after basic combat training in cadets of Indonesia | 12 weeks
  Pre post data in sleep quality using Pittsburgh Sleep Quality Index (psqi) questionnairres consist of 7 component sleep quality. The total score range from 0-21 points
Macronutrient intake before and after basic combat training in cadets of Indonesia | 12 weeks
  Pre post data in total daily intake of carbohydrate,fat, and protein in grams and calories in kilo calorie based on semi quantitave food frequency questionnaires for macronutrient in bahasa Indonesia
Physical activity before and after basic combat training in cadets of Indonesia | 12 weeks
  Pre post data of physical activity in Mets measured by The International Physical Activity Questionnaire (IPAQ) questionairres in bahasa indonesia

CONTACTS AND LOCATIONS:
Locations (1):
- Indonesia Defense University, Bogor, West Java, Indonesia

IPD SHARING:
Plan to Share IPD: No